CLINICAL TRIAL: NCT04946461
Title: Objectifying the Day-time Response Variation of (Lis)Dexamphetamine in Adults With ADHD
Brief Title: The Day-time Response Variation of (Lis)Dexamphetamine
Acronym: IDEAL
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: ADHDcentraal (Unknown)
Responsible Party: Principal Investigator, R.K.R.W. Wettstein, Principal investigator, Amsterdam UMC, location VUmc
Other Study IDs: NL77195.018.21
Record Dates: First submitted 2021-03-30; First posted 2021-06-30 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Adhd
Keywords: Dexamphetamine; lisdexamphetamine; ADHD; QbTest; Pharmacokinetics and dynamics
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Amphetamine; Tablets; Lisdexamfetamine Dimesylate; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A total of 12 blood samples (2 ml per sample) per subject will be taken.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- group 1; lisdex - dex: subjects are assigned to group 1 based on the type of medication prescribed by the practitioner. Subjects which started with lisdexamphetamine are assigned to group 1.
  Interventions: Drug: Dexamfetamine Sulfate 5 Mg Oral Tablet; Drug: Lisdexamfetamine Dimesylate; Biological: blood samples
- group 2; dex - lisdex: subjects are assigned to group 2 based on the type of medication prescribed by the practitioner. Subjects which started with dexamphetamine are assigned to group 1.
  Interventions: Drug: Dexamfetamine Sulfate 5 Mg Oral Tablet; Drug: Lisdexamfetamine Dimesylate; Biological: blood samples

INTERVENTIONS:
Drug: Dexamfetamine Sulfate 5 Mg Oral Tablet — The dosage is set based on the recommendation of the practitioner. Dexamphetamine is administered twice a day, with an interval of 4 hours.
  Other Names: Tentin
Drug: Lisdexamfetamine Dimesylate — The dosage is set based on the recommendation of the practitioner. Lisdexamphetamine is only administered once a day.
  Other Names: Elvanse
Biological: blood samples — The blood samples will be taken at set times: 0, 2, 4, 6, 9 and 12 (hours)
  Other Names: vena puncture

SUMMARY:
In the Netherlands, two forms of amphetamines are available for the treatment of ADHD in adults; dexamfetamine (Tentin) and lisdexamfetamine (Elvanse) and both belong to regular and primary care pharmacotherapy. Both drugs contain exactly the same substance dexamfetamine and it would be expected that the effects on the symptoms of ADHD and the duration of action should be comparable. Previous studies and daily practice have reported different effects and duration of action of both, however. In this study the investigators want to investigate this difference by giving both drugs to the same patient, objectify the blood concentrations, objective and subjective effects and hope to be able to further optimize the treatment for ADHD with amphetamines.

DETAILED DESCRIPTION:
Rationale: In the Netherlands, two types of amphetamines are available for the treatment of adults with ADHD: dexamphetamine sulfate (dex[Tentin ©]) and lisdexamphetamine dimesylate (lisdex [Elvanse ©]) Lisdex is promoted by the manufacturer as a long-acting preparation with a controlled release profile and thus an extended duration of action compared to dex, however, the scientific evidence about the pharmacokinetic (PK) / dynamic (PD) profile of lisdex compared to dex is sparse. Additionally, there are no head-to-head comparisons between dex and lisdex where an objective measurement for the symptom amelioration of ADHD has been used and compared to the plasma concentrations. The hypothesis is that two-times daily dex is more effective in suppressing ADHD symptomatology than once daily lisdex.

Objective: The objective is to compare the pharmacodynamic profile of dex and lisdex in adult patients with ADHD and determine whether the day-time response variation in ADHD symptomatology depends on the type of amphetamine and it's pharmacokinetics.

Study design: An observational study.

Study population: N=16 adults with a minimal age of 18 years old, diagnosed with ADHD according to the DSM 5 criteria, where treatment as usual (TAU) with dex or lisdex already commenced but where the optimal dosage and type of amphetamine have not been established.

Intervention: Sixteen participants will be observed for two consecutive days and PK/PD profiles of lisdex and dex will be observed. Lisdex will be bioequivalently dosed; lisdex once a day and dex two times a day with an interval of 4 hours (TAU). The participants will be observed for approximately 14 hours each day. Blood samples, the Quantified behavior Test (QbTest), physical measurements and questionnaires for drug effects will be taken 6 times at; 0, 2; 4; 6; 9; 12 (hours).

Main study parameters/endpoints: The primary study parameters are the PK/PD profile over time; next to blood samples for pharmacokinetic profiling pharmacodynamic assessments include the QbTest, the drug effect Questionnaire (DEQ), the Bond-Lader Visual Analog Scale (BL-VAS), QbTest performance questionnaire and physical measurements; blood pressure and heart rate.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There are no specific benefits for the study participants. The burden of participating in this study include two extra visits to the outpatient clinic. During each visit the study participant has to fill out some questionnaires, undergo six QbTests and bloodtests. In our opinion the burden for each study participant is considered minor and the risk very low. The therapy given during the study is according to the TAU, which is based on the guidelines of the Dutch association of psychiatry (NVvP) for the treatment of ADHD in adults. The participants will undergo a total of 12 blood samples (2ml per sample). This risk is acceptable in relation to the possible benefits that may be gained from this study, i.e. improved pharmacotherapy guidelines for adult patients with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is aged between 18 - 60 years at time of diagnosis
2. Participant is diagnosed with ADHD according to the DSM 5 criteria
3. Participant started pharmacotherapy treatment with dex or lisdex but no real preference for the type of amphetamine exists according to practitioner
4. Participant is able to provide written informed consent
5. Participant is able and willing to comply with the study protocol

Exclusion Criteria:

1. No diagnosis for ADHD
2. Currently other psychopharmacotherapy treatment than dex or lisdex
3. Currently other psychopharmacotherapy parallel to dex or lisdex

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients who are diagnosed with ADHD according to the DSM 5 criteria (NVvP,2015 ref) at ADHDcentraal and where treatment as usual (TAU) with dex or lisdex already commenced but where the optimal dosage and type of amphetamine has not been established.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Quantified behavior Test (QbTest) | Two consecutive days; the QbTest assessments will be conducted at 6 time points during each day. At baseline (0), repeated after 2, 4, 6, 9 and 12 (hours)
  The pharmacodynamic profile (PD) will be compared to the pharmacokinetic profile to objectify the day-time response variation for both types of amphetamines.
  The QbTest will be used as a PD measure. The QbTest was the world's first FDA cleared, and CE marked ADHD management system. QbTest is a test which objectively evaluates the core symptoms of ADHD for children and adults by combining motion-tracking analysis with a uniquely designed continuous performance task. The test results are compared with an age, length, weight and gender adjusted norm group to set the context to the patient's performance and corresponds to Z-scores (norm population M = 0 and SD =1, SD > 1.5 should be viewed as atypical and give cause for clinical concern).
Drug Effects Questionnaire (DEQ) | Two consecutive days; the DEQ assessments will be conducted at 6 time points during each day. At baseline (0), repeated after 2, 4, 6, 9 and 12 (hours)
  The pharmacodynamic profile (PD) will be compared to the pharmacokinetic profile to objectify the day-time response variation for both types of amphetamines. The DEQ will be used as a PD measure.
  The DEQ is a concise questionnaire, its questions have been widely used and it has shown promising results regarding its psychometric properties. DEQ is therefore suitable for the current study.
  The DEQ consists of 5 items (VAS) that represent the following dimensions: feel of any substance effects (FEEL), feeling of being high (HIGH), drug-liking (LIKE), drug-disliking (DISLIKE) and drug-wanting (MORE). The answers are obtained using a digital VAS scale with numbers that show the values 1 - 100. E.g., A higher score on the LIKE scale represents a higher amount of drug-liking.
Bond-Lader Visual Analog Scale (BL-VAS) | Two consecutive days; the BL-VAS assessments will be conducted at 6 time points during each day. At baseline (0), repeated after 2, 4, 6, 9 and 12 (hours)
  The pharmacodynamic profile (PD) will be compared to the pharmacokinetic profile to objectify the day-time response variation for both types of amphetamines. The BL-VAS will be used as a PD measure.
  The Bond & Lader VAS Mood Rating Scale (BL-VAS) is used to measure the effects of drugs on the participants' mood. The BL-VAS consists of 16 items. The responses are obtained using digital VAS that show the values 1 - 100. The reponses are combined into three dimensions that represent mood, namely: alertness (n = 9), calmness (n = 2) and contentedness (n = 5). The scores of the individual items are summed and averaged, this results in a score for each factor. The range of the factor is 1 - 100. A higher score represents a higher degree of alertness, calmness or contentedness
QbTest performance questionnaire | Two consecutive days; the QbTest performance questionnaire assessments will be conducted at 6 time points during each day. At baseline (0), repeated after 2, 4, 6, 9 and 12 (hours)
  The pharmacodynamic profile (PD) will be compared to the pharmacokinetic profile to objectify the day-time response variation for both types of amphetamines. The QbTest performance questionnaire will be used as a PD measure.
  Participants will perform the QbTest six times a day, immediately after the collection of blood samples. After the QbTest, participants will be shortly questioned about their perception regarding the performance, focus and energy during the test. The questionnaire consists of 4 questions regarding hyperfocus, energy and performance. The responses are obtained using digital VAS that show the values 1 - 100. The scores of the individual items are summed and averaged, this results in a score for each factor. The range of the factor is 1 - 100. A higher score represents a higher degree of performance.
systolic blood pressure (mmHg) | Two consecutive days; the cardiovasculaire assessments will be conducted at 6 time points during each day. At baseline (0), repeated after 2, 4, 6, 9 and 12 (hours)
  The pharmacodynamic profile (PD) will be compared to the pharmacokinetic profile to objectify the day-time response variation for both types of amphetamines. The Cardiovasculaire response will be used as a PD measure.
  Cardiovascular response included blood pressure (diastolic and systolic) and hart rate (puls).
Diastolic blood pressure (mmHg) | Two consecutive days; the cardiovasculaire assessments will be conducted at 6 time points during each day. At baseline (0), repeated after 2, 4, 6, 9 and 12 (hours)
  The pharmacodynamic profile (PD) will be compared to the pharmacokinetic profile to objectify the day-time response variation for both types of amphetamines. The Cardiovasculaire response will be used as a PD measure.
  Cardiovascular response included blood pressure (diastolic and systolic) and hart rate (puls).
Heart rate (heart beats per minute) | Two consecutive days; the cardiovasculaire assessments will be conducted at 6 time points during each day. At baseline (0), repeated after 2, 4, 6, 9 and 12 (hours)
  The pharmacodynamic profile (PD) will be compared to the pharmacokinetic profile to objectify the day-time response variation for both types of amphetamines. The Cardiovasculaire response will be used as a PD measure.
  Cardiovascular response included blood pressure (diastolic and systolic) and heart rate (puls).
Plasma concentration of D-amphetamine | Two consecutive days; the plasma concentration of D-amphetamine will be determined at 6 time points during each day. At baseline (0), repeated after 2, 4, 6, 9 and 12 (hours)
  The PD profiles will be compared to the PK profiles to objectify the day-time response variation for both types of amphetamines. Blood samples, 2ml each, will be collected in lithium heparin tubes 0, 2, 4, 6, 9, 12 h after drug administration. Thereby, the plasma concentration of D-amphetamine can be determined.

SECONDARY OUTCOMES:
Compare area under the curve (AUC) of dex and lisdex | Two consecutive days; blood will be collected at 6 time points during each day. At baseline (0), repeated after 2, 4, 6, 9 and 12 (hours)
  Compare the AUC of dex and lisdex, the investigators hypothesize that the AUC between dex and lisdex will be identical, and the current conversion factor for bioequivalence between dex and lisdex is appropriate.
Compare maximum plasma concentration (Cmax) between lisdex and dex | Two consecutive days; blood will be collected at 6 time points during each day. At baseline (0), repeated after 2, 4, 6, 9 and 12 (hours)
  The investigators hypothesize that the Cmax for lisdex will be higher compared to dex.
Compare time to reach maximum plasma concentration (Tmax) between lisdex and dex | Two consecutive days; blood will be collected at time points: 0, 2, 4, 6, 9 and 12 (hours)
  The investigators hypothesize that Lisdex will have higher drug-liking scores at Tmax than dex.
  The investigators hypothesize that Lisdex will have more side-effects at Tmax than dex.

OTHER OUTCOMES:
The Leeds Sleep Evaluation Questionnaire (LSEQ) | Two consecutive days; the LSEQ will only be conducted at baseline (T0) for each study day
  To see if the quality of sleep prior the observational days has an influence on the QbTest performance Sleep deprivation can negatively impact attention functioning in adults with and without ADHD. Sleep deprived participants performed worse on the QbTest (Dan et al. 2020). The response to the LSEQ will be given using a digital VAS that shows values ranging from 1 -100. The scores are averaged and divided by 10 to give a score for the following chronological domains of sleep: getting to sleep (GTS); question 1 - 3, quality of sleep (QOS); question 4 - 5, awakening following sleep (AFS); questions 6 -7, behavior following awakening (BFW); question 8 - 10. Finally, the score of each domain is added which results in an LSEQ-M global score, ranging from 0 - 100. A higher score for the individual or the global score correlates to a better quality of sleep and/or early morning behavior

CONTACTS AND LOCATIONS:
Overall Officials: R. Mathot, PhD, Principal Investigator — AUMC, location AMC
Locations (1):
- ADHDcentraal, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The IPD can be requested through the official website of ADHDcentraal.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Within 1 year.
Access Criteria: The relevant IPD can be requested through the website of ADHDcentraal.
URL: http://www.adhdcentraal.nl